CLINICAL TRIAL: NCT05931575
Title: Safety, Tolerability and Symptomatic Efficacy of the ROCK-Inhibitor Fasudil in Patients With Parkinson's Disease (ROCK-PD)
Brief Title: Safety, Tolerability and Symptomatic Efficacy of the ROCK-Inhibitor Fasudil in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROCK-PD-0000-LIN-0075-I; 01EN2005 (Other Grant/Funding Number: Bundesministerium für Bildung und Forschung (BMBF))
Record Dates: First submitted 2023-06-12; First posted 2023-07-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-05

CONDITIONS: Idiopathic Parkinson´s Disease
MeSH Terms: interventions — fasudil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention arm (low dose) (Experimental): oral Fasudil solution 88 mg/day (2 x 44 mg)
  Interventions: Drug: Fasudil hydrochloride
- intervention arm (high dose) (Experimental): oral Fasudil solution 44 mg/day (2 x 22 mg)
  Interventions: Drug: Fasudil hydrochloride
- Control intervention arm (placebo) (Placebo Comparator): oral placebo solution 2x/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fasudil hydrochloride — Duration of intervention per patient: 22 days; Application scheme: one dose on day 1, two doses on days 2 - 21, one dose on day 22.
  Other Names: Fasudil hydrochloride (Fasudil)
  Arms: intervention arm (high dose); intervention arm (low dose)
Drug: Placebo — 0.05 ml Quinine dihydrochloride solution (from Quinina Labesfal) in screw flask supplemented with 30 ml Glucose 40% solution from miniplasco directly before use
  Other Names: Quinine dihydrochloride solution
  Arms: Control intervention arm (placebo)

SUMMARY:
The aim of this phase Ila trial is to provide evidence on safety, tolerability and symptomatic efficacy of the ROCK-inhibitor Fasudil in patients with early Parkinson's disease (PD). Fasudil has shown neuroprotective and pro-regenerative effects, modulated microglial activity and attenuated alpha-synuclein aggregation in PD models in vitro and in vivo. It has been licensed in Japan since 1995 for the treatment of vasospasms and has a beneficial safety profile arguing for its repurposing. Up to 15 trial centers in Germany will recruit patients. Blinded trial medication will be prepared and shipped by the University Pharmacy Leipzig. Fasudil in two dosages or placebo will be administered orally twice daily to 75 early PD patients for a total of 3 weeks. Safety, tolerability and symptomatic efficacy endpoints will be assessed up to 4 weeks after end of treatment. Its well-known safety profile and the lack of disease-modifying treatments for PD justifies its use in patients with early Parkinson's disease. ROCK-PD is a prerequisite for subsequent long-term clinical trials assessing disease-modification in PD in addition to symptomatic efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of at least probable PD according to MDS criteria (Postuma et al. MovDis 2015) and
2. Hoehn & Yahr stage 1 - 3
3. must be non-fluctuating (no wearing-off, no dyskinesia) and stable on symptomatic PD medication for at least 6 weeks
4. age: 30 - 80 years
5. Women of childbearing potential must be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test. Acceptable methods of birth control with a low failure rate (i.e. less than 1% per year) when used consistently and correct are for example implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
6. Capable of thoroughly understanding all information given and giving full informed consent according to GCP

Exclusion Criteria:

1. Atypical, secondary Parkinsonian syndromes, PD mimics, or any other medical condition known to have an association with Parkinsonian syndromes, which might confound or obscure the diagnosis of PD
2. Patients with a history of intracranial bleeding, known intracerebral aneurysms or Moyamoya disease, or positive family history for the above. If only family history positive, MR- or x-ray-based cranial imaging not older than 24 months must confirm absence of bleeding, aneurysms, or Moyamoya
3. Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
4. Patients with known arterial hypotension (resting blood pressure <90/60 mmHg) or previous hypotensive episodes or requiring treatment for increasing of blood pressure, such as fludrocortisone, midodrine, etilefrine, cafedrine, or theodrenaline
5. Patients with an uncontrollable or unstable arterial hypertensive disease (resting blood pressure >180 mmHg systolic and/or >120 mmHg diastolic under current antihypertensive medication)
6. Known pulmonary hypertension and any medication prescribed for treatment of pulmonary hypertension
7. Confirmed hepatic insufficiency or abnormal liver function (stable ASAT and/or ALAT greater than 3 times the upper limit of the normal range) and determined to be non-transient through repeat testing
8. Renal insufficiency with a glomerular filtration rate (GFR) <60 ml/min/1,73m² (calculated by MDRD equation or byCKD-EPI equation) and determined to be non-transient through repeat testing
9. Major psychiatric disorder, significant cognitive impairment or clinically evident dementia precluding evaluation of symptoms
10. Hypersensitivity to any component of the IMP
11. Liable to be not cooperative or comply with the trial requirements (as assessed by the investigator), or unable to be reached in the case of emergency
12. Pregnant or breast-feeding females or females with childbearing potential, if no adequate contraceptive measures are used
13. Previous participation in another clinical study involving trial medication within the preceding 12 weeks or five terminal half times of the longest to be eliminated trial medications (whichever is longer) or previous participation in this trial

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Combined occurrence of intolerance and/or occurrence of self-reported and pre-defined treatment-related SAEs | from day 1 to day 22
  Combined occurrence of intolerance (termination of treatment because of treatment-related AE) and/or occurrence of self-reported and pre-defined (laboratory, vital signs) treatment-related SAEs

SECONDARY OUTCOMES:
Occurrence of intolerance | from day 1 to day 22
  Occurrence of intolerance (termination of treatment because of treatment-related AE)
Occurrence of self-reported and pre-defined treatment-related SAEs | from day 1 to day 22, and day 1 to day 50
  Occurrence of self-reported and pre-defined (laboratory, vital signs) treatment-related SAEs
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | part I and II from day 1 to day 22, and day 1 to day 50; time frame: part III and IV from day 1 to day 10, day 1 to day 22, and day 1 to day 50
  the change of MDS-Unified PD Rating Scale (MDS-UPDRS) each part I to IV, min-max: 0-260, 0 indicating no disability and 260 indicating total disability, Part I: Nonmotor experiences of daily living: 13 items. Score range: 0-52; Part II: Motor experiences of daily living: 13 items. Score range: 0-52; Part III: Motor examination: 18 items. Score range: 0-132; Part IV: Motor complications: 6 items. Score range: 0-24; Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe).
MDS-Unified PD Rating Scale (MDS-UPDRS) score | from day 1 to day 22, and day 1 to day 50
  the change of MDS-Unified PD Rating Scale (MDS-UPDRS) score part I to IV, min-max: 0-260, 0 indicating no disability and 260 indicating total disability, Part I: Nonmotor experiences of daily living: 13 items. Score range: 0-52; Part II: Motor experiences of daily living: 13 items. Score range: 0-52; Part III: Motor examination: 18 items. Score range: 0-132; Part IV: Motor complications: 6 items. Score range: 0-24; Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe).
Parkinson's Disease Questionnaire (PDQ-8) | from day 1 to day 22, and day 1 to day 50
  the change of 8-item PD Quality of Life Scale (PDQ-8), min-max: 0-32, 0 no and 32 max
Non-Motor Symptom Questionnaire (NMSQuest) | from day 1 to day 10, day 1 to day 22, and day 1 to day 50
  the change of PD Non-Motor Symptom Questionnaire (NMSQuest), min-max: 0-30, 0 no and 30 max
Montreal Cognitive Assessment (MoCA) | from day 1 to day 22, and day 1 to day 50
  the change of Montreal Cognitive Assessment (MoCA), Montreal Cognitive Assessment MoCA: min-max: 0 (worse) -30 (better outcome)
Beck's Depression Inventory II (BDI-II) | from day 1 to day 22, and day 1 to day 50
  the change of Becks depression inventory-II (BDI-II), min-max: 0-63, 0 no and 63 max
Clinician Global Impression of Improvement (CGI-I) and Patient Global Impression of Improvement (PGI-I) | at day 10, 22 and day 50
  CGI-I [clinician]: min-max: 1-7, min-max: 1 (better) -7 (worse outcome) PGI-I [patient]: min-max: 1-7, min-max: 1 (better) -7 (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lingor, MD, Principal Investigator — Technische Universität München, Klinikum rechts der Isar, Klinik und Poliklinik für Neurologie
Locations (1):
- Technische Universität München, Klinikum rechts der Isar, Klinik und Poliklinik für Neurologie, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolff AW, Bidner H, Remane Y, Zimmer J, Aarsland D, Rascol O, Wyse RK, Hapfelmeier A, Lingor P. Protocol for a randomized, placebo-controlled, double-blind phase IIa study of the safety, tolerability, and symptomatic efficacy of the ROCK-inhibitor Fasudil in patients with Parkinson's disease (ROCK-PD). Front Aging Neurosci. 2024 Feb 14;16:1308577. doi: 10.3389/fnagi.2024.1308577. eCollection 2024. PMID 38419648